CLINICAL TRIAL: NCT04430608
Title: Remote Glucose Monitoring of Patients With Diabetes Quarantined During the COVID-19 Pandemic - a Hospital-Based Randomized Controlled Trial of the Effect of Remote Continuous Glucose Monitoring Compared to Usual Glucose Monitoring
Brief Title: Remote Continues Glucose Monitoring During the COVID-19 Pandemic in Quarantined Hospitalized Patients
Acronym: CGM-ISO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-20025305
Record Dates: First submitted 2020-05-26; First posted 2020-06-12 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2020-05

CONDITIONS: Diabetes; Covid-19; Infection
Keywords: endocrinology; diabetes; quarentine; isolation; CGM
MeSH Terms: conditions — Diabetes Mellitus; COVID-19; Infections

STUDY DESIGN:
Intervention Model Description: Patients are randomized 1:1 to either CGM or Fingerprick group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Fingerprick glucose (Other): Standard care with fingerprick glucose + blinded CGM stratification on COVID-19 status
  Interventions: Device: Dexcom G6
- Open continous glucose monitoring (CGM) (Experimental): Standard care with fingerprick glucose + un-blinded CGM stratification on COVID-19 status
  Interventions: Device: Dexcom G6

INTERVENTIONS:
Device: Dexcom G6 — The investigational device is a CGM Dexcom G6. The Dexcom G6 System is intended to replace fingerstick blood glucose testing for diabetes treatment decisions. The device-system consists of a sensor, the Dexcom G6 device/sender, and connects to a smart device like a cellphone. The Dexcom G6 CGM system is probably the most precise system on the market and with no need for daily calibration with finger prick glucose. The Dexcom G6 sensor can last for 10 days without calibration and is approved for diabetes treatment decision making. Dexcom G6 has been extensively tested and is safe and approved even for pregnant women.
  The CE Marking confirms that the G6 system meets the Essential Requirements of the Medical Device Directive MDD 93/42/EEC as amended by 2007/47/EC.

SUMMARY:
This is a randomized controlled trial of isolated patients with diabetes admitted to Nordsjællands Hospital with or without COVID-19-pneumonia. A continuous glucose monitoring (CGM) based system with transmission of glucose data to a central system is used for remote monitoring of glucose levels and compared to standard finger-prick glucose. Blinded (to patients) CGM is mounted in the finger-prick group.

DETAILED DESCRIPTION:
Epidemics and pandemics are a constant threat to health care systems globally. This stresses the importance of preparedness for a large amount of hospitalized quarantined patients in isolation, with the extra challenges it brings. The COVID-19 pandemic challenges the Danish health care system in many aspects: An increased number of citizens are expected to be admitted to hospital due to COVID-19 infected pneumonia and this will demand extra workforce resources, extra use of protective equipment (gowns, masks, gloves, etc) and extra time used for taking protective equipment on and off. In concert these extra demands will drain the health care system and any initiative to reduce these challenges is needed.

In this randomized controlled trial, isolated patients with diabetes will be randomized to either standard care fingerprick glucose + blinded CGM or Dexcom G6 only.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized with confirmed COVID-19 infection by real-time PCR or another validated method OR hospitalized with a non-COVID-19 diagnosis AND in isolation at time of inclusion.
2. A documented clinically relevant history of diabetes or newly discovered during hospitalization.
3. Written informed consent obtained before any trial related procedures are performed.
4. Male or female aged over 18 years of age.
5. Must be able to communicate with the study personnel.
6. The subject must be willing and able to comply with trial protocol.

Exclusion Criteria:

1. Known hypersensitivity to the band-aid of the Dexcom G6 sensors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-04-25 (Actual)

PRIMARY OUTCOMES:
Time In Range (TIR) for blood glucose | 1-2 weeks
  TIR is presented in percent of time in which the participants' glucose values are in different glucose ranges.

SECONDARY OUTCOMES:
Saved patient-personnel contacts related to blood glucose measurements. | 1-2 weeks
  Saved patient-personnel contacts related to blood glucose measurements, incl. time healthcare providers spent on diabetes related tasks and PPE related tasks, during the patients' hospitalization.
Glucose variations during hospitalization | 1-2 weeks
  Additional glucose outcomes based on data from Dexcom G6 are for example Time Above Range (TAR), Time Below Range (TBR), average glucose, variance in glucose (CV), etc.
Blood glucose lowering interventions | 1-2 weeks
  That is: Tablet-based and insulin-based regimens and number of times that sliding scale insulin (including dose of insulin) has been administered for each patient.
CGM sensor performance | 1-2 weeks
  Number of techincal errors during the sensors lifetime.
Course of hospital stay. | 1-2 weeks
  Hospital death (yes/no), length of stay at hospital, need for respiratory support (yes/no) and intensive care (yes/no), recovered vs. fatal (death within 60 days from admission).

CONTACTS AND LOCATIONS:
Overall Officials: Peter L. Kristensen, MD, ph.D, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Nordsjællands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No
Undecided, will be updated

REFERENCES:
- [Derived] Klarskov CK, Windum NA, Olsen MT, Dungu AM, Jensen AK, Lindegaard B, Pedersen-Bjergaard U, Kristensen PL. Telemetric Continuous Glucose Monitoring During the COVID-19 Pandemic in Isolated Hospitalized Patients in Denmark: A Randomized Controlled Exploratory Trial. Diabetes Technol Ther. 2022 Feb;24(2):102-112. doi: 10.1089/dia.2021.0291. Epub 2022 Jan 4. PMID 34524009
- [Derived] Klarskov CK, Lindegaard B, Pedersen-Bjergaard U, Kristensen PL. Remote continuous glucose monitoring during the COVID-19 pandemic in quarantined hospitalized patients in Denmark: A structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Nov 25;21(1):968. doi: 10.1186/s13063-020-04872-4. PMID 33239100